CLINICAL TRIAL: NCT02919280
Title: Dallas 2K: A Natural History Study of Depression
Acronym: D2K
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The Hersh Foundation (Unknown)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 112015-021
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Depression; Depression, Bipolar
Keywords: healthy control; depression; bipolar
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Establish a D2K biospecimen resource consisting of stool, blood, plasma, serum, PBMCs, buffy coat, RNA, and saliva collected from participants at baseline and at follow-up visits, as a platform for translational research into biochemical and molecular characterization of depression.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: This is an observational study. No intervention / treatment involved.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — The Dallas 2K is a 10-year natural history, longitudinal, prospective study of a cohort of 2,500 participants. There is no medication or non-medication treatment or intervention provided by this study.

SUMMARY:
The primary objective of this initiative is to implement a prospective study that will allow us to identify and validate biosignatures of response to treatments for depression and depression outcome (using an integrated array of participant specific data: socio-demographic, lifestyle, clinical and behavioral assessments, fluid-based biomarkers, genomics, neuroimaging, EEG, and cell-based assays) in a longitudinal cohort of subjects with elevated symptoms of a depressive disorder.

Symptom remission across various treatment options will be assessed using questionnaires for symptom changes, antidepressant treatment tolerability and overall quality of life. Other outcomes generated from this study will include rate of change in quantitative measures of brain function, of depression relevant brain regions correlated with systems-levels behavior and other functional neuro-circuitry MRI measures. Rate of change of specified biochemical biomarkers will also be assessed.

Integration of these measures will provide an unmatched understanding into the mechanisms of depression and hold tremendous promise for better disease treatment and associated outcomes.

DETAILED DESCRIPTION:
D2K is a 10-year natural history, longitudinal, prospective study of a cohort of 2,500 participants that will help uncover the socio-demographic, lifestyle, clinical, psychological, and neurobiological factors that contribute to antidepressant treatment response: remission, recurrence, relapse and individual outcomes in depressive disorders. As this is an exploratory study, we will assess a comprehensive panel of carefully selected participant specific parameters: socio-demographic (age, sex, gender, race, ethnicity, economic); life habits (physical activity, substance use); clinical (medical history, anxious depression, early life trauma), biological (biomarkers in blood, saliva, urine, stool), behavioral (cognitive, emotional), neurophysiological (EEG), and neuroimaging (magnetic resonance imaging; MRI) with the goal of developing the most robust predictive models of depression treatment response and of outcomes.

Clinician rated assessments, participant rated assessments, blood, saliva, stool, and urine collection, EEG, and MRI will be performed during the duration of the study. An optional m-health study may be collected continuously via a phone application and/or wristband over the course of the study. With this said, due to the nature of the protocol and the large number of research participants, we expect some appointments that include procedures and assessments to be missed within an expected study time frame. We will attempt to complete any missed appointments at the next scheduled visit. For the purposes of this study, missed procedures and/or assessments are not considered protocol deviations. In addition, the schedule of assessments to be completed will vary from time to time within this longitudinal study to help balance the data between age, sex, biological gender, gender identity, sexual orientation, gender expression, and diagnosis breakdown of our enrolled participants for data analyses.

The schedule of assessments will NOT exceed the following:

1. Monthly Surveys: 12 times a year
2. MRI: up to 4 times a year
3. EEG: up to 4 times a year
4. Biospecimen collection: up to 4 times a year
5. Cognitive Behavioral Tasks: up to 4 times a year
6. Extensive Self-report and Clinician rated assessments: 4 times a year
7. Stool Sample collection: up to 4 times a year
8. Optional M-health: Duration of the study (starting from Baseline) Participants will be compensated based on the study activity they complete and will not exceed the total amount (per year) that is approved by the IRB. No study procedures will be conducted until signed informed consent has been obtained from the participant. Details regarding informed consent procedures are included in section 8.

Procedures specific to youth 17 years old or younger: Participants will complete the questionnaires that have been normed and validated to their age with the assistance of study staff. Forms may also be completed by participant's parent(s)/guardian(s)/LAR as needed.

ELIGIBILITY:
Criteria for Inclusion of participants:

A potential participant will be eligible for participation in this study if the following criteria are met:

1. Male and female adult or youth aged 10 and older of any race or ethnicity.
2. Ability to speak, read, and understand English. However, the parent(s) or legal guardians of minors may either speak English or Spanish as the consenting process can be conducted bilingually.
3. A lifetime or a current diagnosis of a mood disorder based upon a semi-structured diagnostic interview.
4. Adults age 18 and older must be able to provide written informed consent; for youth younger than age 18, a parent or legal guardian must provide written informed consent, and the child or teen must provide written informed assent.

Eligibility for Healthy Controls

For comparison purposes, potential health control participants who do NOT have a psychiatric diagnosis will be enrolled as part of the healthy control arm of this study.

1. Male and female adult or youth aged 10 and older of any race or ethnicity.
2. Ability to speak, read, and understand English. However, the parent(s) or legal guardians of minors may either speak English or Spanish as the consenting process can be conducted bilingually.
3. Adults age 18 and older must be able to provide written informed consent; for youth younger than age 18, a parent or legal guardian must provide written informed consent, and the child or teen must provide written informed assent.

Criteria for Exclusion of Participants

A potential participant will NOT be eligible for participation in this study if any of the following criteria are met:

1. History of schizophrenia, schizoaffective disorders or chronic psychotic disorders based upon a semi-structured diagnostic interview.
2. Diagnosis of human immunodeficiency virus (HIV) or hepatitis B or C (human immunodeficiency virus (HIV) testing is not required for this study).
3. Unable to provide a stable home address and contact information.
4. Has any condition for which, in the opinion of the investigator or designee, study participation would not be in their best interest (including but not limited to cognitive impairment, unstable general medical condition, intoxication, active psychosis) or that could prevent, limit, or confound the protocol-specified assessments.
5. Requires immediate hospitalization for psychiatric disorder or suicidal risk as assessed by a licensed study clinician.

Eligibility for Healthy Controls

A potential Healthy Control participant will NOT be eligible for participation in this study if any of the following criteria are met:

1. A lifetime or a current history of a mood disorder based upon a semi-structured diagnostic interview.
2. Meets any exclusion criteria as part of the main D2K study interview.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The following group is being targeted for this observational study:
  1. Depressed patients
  2. Lifetime or Current Diagnosis of a Mood Disorder
  3. Bipolar Disorder
  4. Health Controls with NO Psychiatric Diagnosis ( For Comparison Purposes)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-06-14 (Actual); Primary Completion 2036-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes in depression severity of subjects with elevated symptomatology on Patient Health Questionnaire (PHQ-9) for non-psychotic depressive disorders. | 10 years

SECONDARY OUTCOMES:
Comparison of Longitudinal changes in functioning as measured by Magnetic Resonance imaging in patients with severe depression | 10 years
Comparison of Longitudinal changes in functioning as measured by quantitative electroencephalography (EEG) in patients with severe depression. | 10 years
Comparison of Longitudinal changes in fluid based biomarkers as measured by proteomic methods in patients with severe depression. | 10 years
Comparison of Longitudinal changes in fluid based biomarkers as measured by metabolomics methods in patients with severe depression. | 10 years
Comparison of Longitudinal changes in fluid based biomarkers as measured by transcriptomic methods in patients with severe depression. | 10 years
Comparison of Longitudinal changes in fluid based biomarkers as measured by genomic methods in patients with severe depression. | 10 years
Comparison of Longitudinal changes in fluid based biomarkers as measured by epigenomic methods in patients with severe depression. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Result] Trivedi MH, Greer TL, Grannemann BD, Church TS, Somoza E, Blair SN, Szapocznik J, Stoutenberg M, Rethorst C, Warden D, Ring KM, Walker R, Morris DW, Kosinski AS, Kyle T, Marcus B, Crowell B, Oden N, Nunes E. Stimulant reduction intervention using dosed exercise (STRIDE) - CTN 0037: study protocol for a randomized controlled trial. Trials. 2011 Sep 19;12:206. doi: 10.1186/1745-6215-12-206. PMID 21929768
- [Result] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Result] Bloom BS. Prevalence and economic effects of depression. Manag Care. 2004 Jun;13(6 Suppl Depression):9-16. PMID 15293766
- [Derived] Chin Fatt CR, Minhajuddin A, Goodman LC, Vasu S, Mayes TL, Sethuram S, Trombello JM, Hughes JL, Greer TL, Foster JA, Trivedi MH. Defining anhedonia subgroups using the dimensional anhedonia rating scale in active depression: Findings from the Texas resilience against depression study. J Psychiatr Res. 2026 Feb;193:480-486. doi: 10.1016/j.jpsychires.2025.12.023. Epub 2025 Dec 11. PMID 41401669